CLINICAL TRIAL: NCT00593762
Title: Investigation of Laboratory Resistance to Aspirin and Clopidogrel and Its Clinical Relevance in Patients With Peripheral Arterial Occlusive Disease Requiring Interventional Procedures
Brief Title: ASA- and Clopidogrel-Responsiveness in Patients With Peripheral Arterial Occlusive Disease and Interventional Procedures
Status: Suspended | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: PD Dr. E. Lindhoff-Last, Division of Vascular Medicine, Department of Internal Medicine, J.W.Goethe University Hospital Frankfurt
Other Study IDs: E 19/05
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2008-01

CONDITIONS: Peripheral Arterial Occlusive Disease
Keywords: Peripheral arterial occlusive disease; Aspirin; Clopidogrel; Resistance; Catheter interventional procedure; ASA and clopidogrel resistance
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to determine the response to aspirin (ASA) and Clopidogrel in patients with peripheral arterial occlusive disease (PAOD) requiring interventional procedures and to investigate if patients with "resistance" to ASA or Clopidogrel have an unfavourable outcome during long-term follow-up

ELIGIBILITY:
Inclusion Criteria:

* PAOD patients
* Age 18-85 years
* Need for a catheter interventional procedure
* Antithrombotic therapy with aspirin or clopidogrel

Exclusion Criteria:

* Comedication additionally compromising platelet function
* Known bleeding disorder
* Life expectancy < 6 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with peripheral arterial occlusive disease (PAOD) requiring a catheter interventional procedure
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2005-05; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Need for peripheral arterial revascularisation | 1, 6, 12 and 24 months

SECONDARY OUTCOMES:
Cardiovascular events (death, myocardial infarction, stroke, ACS, PCI) | 1, 6, 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Linnemann, MD, Principal Investigator — Division of Vascular Medicine, Department of Internal Medicine, J.W. Goethe University Hospital Frankfurt
Locations (1):
- Division of Vascular Medicine, Department of Internal Medicine, J.W.Goethe University Hospital, Frankfurt am Main, Hesse, Germany